CLINICAL TRIAL: NCT04756544
Title: he Influence of Probiotic Supplementation on Depressive Symptoms, Inflammation and Oxidative Stress Parameters and Faecal Microbiota in Patients With Depression Depending on Metabolic Syndrome Comorbidity
Brief Title: The Influence of Probiotic Supplementation on Depressive Symptoms, Inflammation and Oxidative Stress Parameters and Faecal Microbiota in Patients With Depression Depending on Metabolic Syndrome Comorbidity
Acronym: PRO-DEMET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Oliwia Gawlik-Kotelnicka, MD, PhD, Dr., Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RNN/228/20/KE
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Depressive Disorder; Depression; Anxiety; Stress; Metabolic Syndrome; NAFLD
Keywords: depression; metabolic syndrome; probiotics; microbiota; inflammation; oxidative stress
MeSH Terms: conditions — Depressive Disorder; Depression; Anxiety Disorders; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Depressive Disorders + probiotic (Experimental)
  Interventions: Dietary Supplement: Lactobacillus helveticus Rosell®-52, Bifidobacterium longum Rosell®-175
- Depressive Disorders + placebo (Placebo Comparator)
  Interventions: Other: placebo
- Depressive disorder + metabolic syndrome + probiotic (Experimental)
  Interventions: Dietary Supplement: Lactobacillus helveticus Rosell®-52, Bifidobacterium longum Rosell®-175
- Depressive disorder + metabolic syndrome + placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus helveticus Rosell®-52, Bifidobacterium longum Rosell®-175 — probiotic
  Arms: Depressive Disorders + probiotic; Depressive disorder + metabolic syndrome + probiotic
Other: placebo — placebo
  Arms: Depressive Disorders + placebo; Depressive disorder + metabolic syndrome + placebo

SUMMARY:
The trial will be a four-arm, parallel group, prospective, randomized, double-blind, controlled design that will include 200 participants and will last 20 weeks. The probiotic preparation will contain Lactobacillus helveticus Rosell®-52, Bifidobacterium longum Rosell®-175. We will assess the level of depression, anxiety and stress, quality of life, blood pressure, body mass index and waist circumference, white blood cells count, serum levels of C-reactive protein, HDL cholesterol, triglicerides, fasting glucose, faecal microbiota composition and the level of some faecal microbiota metabolites, as well as inflammation markers and oxidative stress parameters in serum.

The trial may establish a safe and easy-to-use treatment option as an adjunct in a subpopulation of depressive patients only partially responsive to pharmacologic treatment.

ELIGIBILITY:
Inclusion Criteria:

Depressive disorders diagnosed according to ICD Age between 18 and 70 years MADRS score >=13 Antidepressant and antianxiety medications or psychotherapy not changed 3 weeks prior to the beginning of the study DMS study groups: MetS diagnosed according to International Diabetes Federation (IDF)

Exclusion Criteria:

Pregnancy; An infection and/or treatment with antibiotics in the previous 4 weeks; Supplementation with pro- or prebiotics in the previous 4 weeks; Having a diagnosis of autoimmune, serious immunocompromised, inflammatory bowel diseases, cancer, IgE-dependent allergy, severe kidney failure or unstable thyroid dysfunction in the previous 4 weeks; Psychiatric comorbidities (except for specific personality disorder, additional specific anxiety disorder and caffeine or nicotine addiction); Regular treatment (more than 3 days a week) with proton-pump inhibitors (PPIs), metformin, laxatives, systemic steroids or nonsteroidal anti-inflammatory drugs (NSAIDs) in the previous 4 weeks; Following a specific diet or a significant change in dietary pattern in the previous 4 weeks; Significant change in daily physical activity or an extreme sport activity in the previous 4 weeks; Significant change in dietary supplementation in the previous 4 weeks; Significant change in smoking pattern in the previous 4 weeks; A major neurological disorder or any medical disability that may interfere with a subject's ability to complete study procedures; High risk of suicide according to Tool of Assessment of Suicide Risk (TASR); Is participating in, or has recently participated in, another research study involving an intervention which may alter outcomes of interest to this study; Any other condition or situation which, in the view of investigators, would affect the compliance or safety of the individual taking part; D study groups: MetS diagnosed according to International Diabetes Federation (IDF).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
depressive symptoms | 2 years
  MADRS score

CONTACTS AND LOCATIONS:
Locations (1):
- Oliwia Gawlik-Kotelnicka, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kotelnicka OG, Wysokinski A, Gajewska A, Czarnecka-Chrebelska K, Kopacz K, Skowronska A, Pikus E, Brzezianska-Lasota E, Strzelecki D. Probiotics Decrease C-Reactive Protein Levels in Depression Depending on Metabolic Syndrome Presence or Antidepressant Treatment - Secondary Results of a Randomized Clinical Trial. Curr Neuropharmacol. 2025 Oct 29. doi: 10.2174/011570159X371175251002220658. Online ahead of print. PMID 41177800
- [Derived] Gawlik-Kotelnicka O, Sobczak M, Palma J, Poplawska M, Skonieczna-Zydecka K, Plewka M, Pawliczak R, Strzelecki D. Does isovaleric acid play a key role in the interaction between probiotics and antidepressants? A secondary analysis of a randomized clinical trial. Comput Struct Biotechnol J. 2025 May 27;27:2275-2287. doi: 10.1016/j.csbj.2025.05.035. eCollection 2025. PMID 40520599
- [Derived] Gawlik-Kotelnicka O, Rogalski J, Czarnecka-Chrebelska KH, Burzynski J, Jakubowska P, Skowronska A, Strzelecki D. The Interplay Between Depression, Probiotics, Diet, Immunometabolic Health, the Gut, and the Liver-A Secondary Analysis of the Pro-Demet Randomized Clinical Trial. Nutrients. 2024 Nov 24;16(23):4024. doi: 10.3390/nu16234024. PMID 39683419
- [Derived] Gawlik-Kotelnicka O, Burzynski J, Rogalski J, Skowronska A, Strzelecki D. Probiotics may be useful for drug-induced liver dysfunction in patients with depression - A secondary analysis of a randomized clinical trial. Clin Nutr ESPEN. 2024 Oct;63:604-614. doi: 10.1016/j.clnesp.2024.07.1024. Epub 2024 Jul 30. PMID 39089652
- [Derived] Gawlik-Kotelnicka O, Margulska A, Pleska K, Skowronska A, Strzelecki D. Metabolic Status Influences Probiotic Efficacy for Depression-PRO-DEMET Randomized Clinical Trial Results. Nutrients. 2024 May 3;16(9):1389. doi: 10.3390/nu16091389. PMID 38732635
- [Derived] Gawlik-Kotelnicka O, Skowronska A, Margulska A, Czarnecka-Chrebelska KH, Loniewski I, Skonieczna-Zydecka K, Strzelecki D. The Influence of Probiotic Supplementation on Depressive Symptoms, Inflammation, and Oxidative Stress Parameters and Fecal Microbiota in Patients with Depression Depending on Metabolic Syndrome Comorbidity-PRO-DEMET Randomized Study Protocol. J Clin Med. 2021 Mar 24;10(7):1342. doi: 10.3390/jcm10071342. PMID 33804999